CLINICAL TRIAL: NCT03586609
Title: Phase II Study of Venetoclax Added to Cladribine Plus Low Dose Cytarabine (LDAC) Induction Followed by Consolidation With Cladribine Plus LDAC Alternating With 5-Azacitidine With Venetoclax in Patients With Untreated AML
Brief Title: Venetoclax, Cladribine, Low Dose Cytarabine, and Azacitidine in Treating Patients With Previously Untreated Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0020; NCI-2018-01318 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0020 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Cladribine; Cytarabine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cladribine, cytarabine, venetoclax, azacitidine) (Experimental): See Detailed Description.
  Interventions: Drug: Azacitidine; Drug: Cladribine; Drug: Cytarabine; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; Onureg; U-18496; Vidaza
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Cytarabine — Given SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies how well venetoclax, cladribine, low dose cytarabine, and azacitidine work in treating patients with acute myeloid leukemia that has previously not been treated. Drugs used in chemotherapy, such as venetoclax, cladribine, and low dose cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Azacitidine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving venetoclax, cladribine, low dose cytarabine induction followed by cladribine, low dose cytarabine, and azacitidine consolidation may work better in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the complete response (CR/complete response with incomplete recovery [CRi]) rate of patients with acute myeloid leukemia (AML) treated with venetoclax combined with cladribine (2-CDA) plus low-dose cytarabine (LDAC) alternating with 5-azacytidine.

SECONDARY OBJECTIVES:

I. To assess overall survival (OS) of patients with AML treated with venetoclax added to cladribine plus LDAC alternating with 5-azacytidine.

II. To assess the disease free survival (DFS) patients with AML treated with venetoclax added to cladribine plus LDAC alternating with 5-azacytidine and achieved a complete response (CR/CRi).

III. To assess the overall response rate of patients with AML treated with venetoclax added to cladribine plus LDAC alternating with 5-azacytidine.

IV. To assess toxicity and induction mortality of patients with AML treated with venetoclax added to cladribine plus LDAC alternating with 5-azacytidine.

EXPLORATORY OBJECTIVES:

I. Evaluate and determine venetoclax pharmacokinetics (pK) in presence or absence of concomitantly administered drugs such as posaconazole, voriconazole, isafuconazole, and fluconazole.

II. Investigate the correlation between venetoclax pK with toxicities and efficacy.

III. Investigate the correlation of baseline cytogenetic and mutational data with likelihood of response and resistance to the regimen.

IV. Evaluate the depth of response with minimal residual disease (MRD) testing and correlate with long term outcome.

OUTLINE:

INDUCTION: Patients receive cladribine intravenously (IV) daily over 1-2 hours on days 1-5, cytarabine subcutaneously (SC) twice daily (BID) on days 1-10, and venetoclax orally (PO) daily on days 1-21. Treatment continues for 28 days in the absence of disease progression or unacceptable toxicity. Patients who do not achieve a CR or CRi after cycle 1 may receive a second induction cycle. Patients who do not achieve CR or CRi after second induction cycle may proceed to cycle 3 of consolidation per investigator.

CONSOLIDATION/MAINTENANCE:

Patients who achieve CR or CRi after cycle 1 of induction receive cladribine IV over 1-2 hours daily on days 1-3, cytarabine SC BID on days 1-10, and venetoclax PO once daily (QD) on days 1-21 of cycle 2. All patients receive cladribine IV daily over 1-2 hours of cycles 5-6, 9-10, 13-14, and 17-18, cytarabine SC BID on days 1-3 of cycles 5-6, 9-10, 13-14, and 17-18, venetoclax PO QD on days 1-21 of cycle 3-18, and azacitidine SC daily or IV over 30-60 minutes on days 1-7 of cycles 3-4, 7-8, 1-12, and 15-18. Treatment repeats every 28 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-12 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with previously untreated acute myeloid leukemia (AML). Prior therapy with hydroxyurea, hematopoietic growth factors, HMA, ATRA, or a total dose of cytarabine up to 2g (for emergency use for stabilization) is allowed.
2. Age >/= 50 years. Participants aged < 50 years who are unsuitable for standard induction therapy may be eligible after discussion with primary investigator
3. Adequate organ function as defined below:

   * liver function (bilirubin < 2mg/dL, AST and/or ALT <3 x ULN). Unless liver enzyme abnormalities are determined by the treating MD and PI to be due to leukemic infiltration.
   * kidney function (creatinine < 1.5 x ULN ).
4. ECOG performance status of ≤ 2.
5. A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.
6. Participants must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the participants is required prior to their enrollment on the protocol.

Exclusion Criteria:

1. Pregnant women are excluded from this study because the agents used in this study have the potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding should also be avoided.
2. Uncontrolled intercurrent illness including, but not limited to ongoing or active uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Participants with documented hypersensitivity to any of the components of the chemotherapy program.
4. Men and women of childbearing potential who do not practice contraception. Women of childbearing potential and men must agree to use contraception prior to study entry and for the duration of study participation.
5. Prior therapy with venetoclax
6. Participants with a diagnosis of acute promyelocytic leukemia (AML-M3) will be excluded from this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2018-10-25 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of complete response (CR/complete response with incomplete recovery [CRi]) | Up to completion of cycle 2 (each cycle is 28 days)
  The optimum two-stage design will be implemented. Will be estimated along with the 95% confidence intervals.

SECONDARY OUTCOMES:
Overall response rate | Up to 5 years
  Will be estimated along with the 95% confidence intervals.
Overall survival (OS) | Time interval between treatment start and the date of death or last follow-up, whichever occurred first, assessed up to 5 years
  Kaplan-Meier method will be used to assess the OS probabilities. The median OS will be reported, along with the 95% confidence intervals.
Disease-free survival (DFS) | Time interval between treatment start and the date of death or last follow-up, whichever occurred first, assessed up to 5 years
  Kaplan-Meier method will be used to assess the DFS probabilities. The median DFS will be reported, along with the 95% confidence intervals.
Incidence of adverse events graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 5 years
  The Bayesian approach will be implemented for toxicity monitoring, where toxicity is defined as any grade 3 or higher non-hematological toxicity which is at least possibly related to the treatment that occurs during the first 2 cycles of treatment. Safety data will be summarized by category, severity and frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan M Kadia, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kadia TM, Reville PK, Wang X, Rausch CR, Borthakur G, Pemmaraju N, Daver NG, DiNardo CD, Sasaki K, Issa GC, Ohanian M, Montalban-Bravo G, Short NJ, Jain N, Ferrajoli A, Bhalla KN, Jabbour E, Takahashi K, Malla R, Quagliato K, Kanagal-Shamanna R, Popat UR, Andreeff M, Garcia-Manero G, Konopleva MY, Ravandi F, Kantarjian HM. Phase II Study of Venetoclax Added to Cladribine Plus Low-Dose Cytarabine Alternating With 5-Azacitidine in Older Patients With Newly Diagnosed Acute Myeloid Leukemia. J Clin Oncol. 2022 Nov 20;40(33):3848-3857. doi: 10.1200/JCO.21.02823. Epub 2022 Jun 15. PMID 35704787
- See also: MD Anderson Cancer Center — http://www.mdanderson.org